CLINICAL TRIAL: NCT00978523
Title: A Phase 1 Study of AR-12 (2-Amino-N-[4-[5-(2 Phenanthrenyl)-3-(Trifluoromethyl)-1H-pyrazol-1-yl] Phenyl]-Acetamide) in Adult Patients With Advanced or Recurrent Solid Tumors or Lymphoma, for Which No Standard Therapy Is Available
Brief Title: Study of AR-12 (2-Amino-N-[4-[5-(2 Phenanthrenyl)-3-(Trifluoromethyl)-1H-pyrazol-1-yl] Phenyl]-Acetamide) in Adult Patients With Advanced or Recurrent Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arno Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARN-AR12-CT101
Record Dates: First submitted 2009-09-15; First posted 2009-09-17 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Solid Tumors; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — OSU 03012

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with AR-12 (Experimental): This is a single-agent, open-label, Phase 1, dose-escalation study in adult patients with advanced or recurrent solid tumors or lymphoma. Patients will receive orally administered AR-12 once daily for 28 consecutive days. The first dosing cycle will be followed by at least a 7 day off-treatment period; however, no off-treatment period will be scheduled between subsequent treatment cycles
  Interventions: Drug: AR-12: (2-Amino-N-[4-[5-(2 phenanthrenyl)-3-(trifluoromethyl)-1H-pyrazol-1-yl] phenyl]-acetamide)

INTERVENTIONS:
Drug: AR-12: (2-Amino-N-[4-[5-(2 phenanthrenyl)-3-(trifluoromethyl)-1H-pyrazol-1-yl] phenyl]-acetamide) — Oral, dose-escalation

SUMMARY:
The primary objective of this study in adults with advanced or recurrent solid tumors or lymphoma is to evaluate the safety and tolerability of AR-12 by describing dose-limiting toxicities (DLTs), and thereby establishing the maximum tolerated dose (MTD) or, in the absence of reaching an MTD, a recommended dose (RD) for additional study of oral AR-12 administered daily in cycles of 28 days (28 consecutive days of once daily treatment with at least a 7-day break between the first and second treatment cycles and recovery of toxicity to grade 1 or less, with no planned off-treatment days between subsequent cycles).

DETAILED DESCRIPTION:
This is a single-agent, open-label, Phase 1, dose-escalation study in adult patients with advanced or recurrent solid tumors or lymphoma. Patients will receive orally administered AR-12 once daily for 28 consecutive days. The first dosing cycle will be followed by at least a 7 day off-treatment period; however, no off-treatment period will be scheduled between subsequent treatment cycles. If daily dosing is not tolerated by the study population, alternative dosing schedules may be pursued (eg, 21 consecutive days of dosing followed by 7 days off treatment), as indicated by the safety, pharmacokinetic, and pharmacodynamic data; all changes to the protocol-specified dosing schedule must be agreed upon by the investigators and the medical monitor. If individual patients respond to AR-12 treatment with an objective response or stable disease according to RECIST criteria and meet pre-specified retreatment criteria, they may continue to receive cycles of AR-12 in the absence of untoward or serious toxicity; however, no patient is permitted to start a subsequent cycle after each bi-monthly disease evaluation until it is confirmed that disease progression has not occurred.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, written informed consent must be obtained and documented according to International Conference on Harmonisation (ICH) Good Clinical Practice (GCP), the local regulatory requirements, and the permission to use private health information in accordance with the Health Insurance Portability and Accountability Act (HIPAA) prior to study-specific Screening procedures.
2. Both men and women and members of all races and ethnic groups are eligible for this trial.
3. Patients must be 18 years of age or greater.
4. Patients must have a histologically or cytologically confirmed advanced or recurrent solid tumor or lymphoma for which standard curative or palliative measures do not exist or are no longer effective. Patients who have recurrent disease after previous surgery, radiation therapy, and/or chemotherapy are eligible. No restriction is placed on the number of prior therapies. At least 4 weeks must have elapsed since the completion of prior therapy, including major surgery, and patients must have recovered from all associated toxicities no greater than grade 1 at the time of Screening. Patients with prostate cancer must have discontinued anti-androgens (eg, bicalutamide, nilutamide) for at least 6 weeks; chemical castration with LHRH analogues can be continued.
5. Patients must have measurable or evaluable disease or disease that otherwise meets criteria for treatment and can be followed by an acceptable biomarker (eg, PSA or CA-125) documented within 28 days of starting treatment with AR-12. Pleural effusions, ascites, bony metastasis, and laboratory parameters are not acceptable as the only evidence of disease.
6. Patients must have acceptable organ and marrow function documented within 7 days of registration, defined as follows:

   * Leukocytes >3,000/mcL
   * Absolute neutrophil count >1,500/mcL
   * Platelets ≥150,000/mcL
   * Fasting blood glucose Within normal institutional limits
   * Total bilirubin Within normal institutional limits
   * AST/ALT <2.5 X institutional ULN; <5 X ULN in presence of liver metastasis
   * Creatinine Within normal institutional limits, OR
   * Creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
7. Patients must have an ECOG performance status of 0 or 1.
8. Patients must have adequate pulmonary function (no more than a grade 2 finding per CTCAE version 3) and oxygen saturation ≥93% on room air, measured within 14 days prior to initiation of treatment with AR-12.
9. All patients who are sexually active must use a medically acceptable, as judged by the investigator, and highly effective method of birth control for the duration of the study and to continue for 30 days after the last AR-12 dose. A highly effective method of birth control is defined as any method that results in a low failure rate, including implants, injectables, some intrauterine devices, sexual abstinence, and surgical sterilization (eg, vasectomy, tubal ligation, hysterectomy). Women of childbearing potential must have a negative serum pregnancy test documented within 7 days prior to Day 0. Furthermore, male study patients must also not donate sperm from Study Day 1 until 90 days after the end of treatment.
10. Patients must have a life expectancy of greater than 12 weeks.

Exclusion Criteria:

1. Patients must not have had chemotherapy, radiotherapy, immunotherapy, or investigational agents within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study. Patients who have received prior chemotherapy must have recovered to no greater than grade 1 from all AEs/toxicities (except alopecia) due to prior agents.
2. Patients with a history of insulin- or non-insulin-dependent diabetes requiring antidiabetic medication.
3. Patients requiring treatment with anticoagulants.
4. Patients requiring chronic corticosteroids (dose equivalent ≥20 mg prednisolone).
5. Patients requiring chronic Celebrex® (celecoxib) therapy.
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition (eg, celecoxib).
7. Patients who are unable or unwilling to swallow AR-12 capsules daily or who have any concurrent medical condition that may impact drug absorption, including a history suggestive of intermittent tumor-associated bowel obstruction, and partial small bowel resection.
8. Patients with known or symptomatic brain metastases (including leptomeningeal disease). Patients with asymptomatic, treated brain metastases are allowed. Patients with primary brain tumors will be allowed in the MTD expansion cohort; however, radiotherapy must have been completed ≥90 days prior to Screening.
9. Patients with any other prior malignancy are not allowed except for the following:

   * Adequately treated basal cell or squamous cell skin cancer
   * In situ cervical cancer
   * Adequately treated Stage I or II cancer from which the patient is currently in complete remission or other cancer from which the patient has been disease-free for 2 years
10. Patients may have had prior palliative radiation therapy; however, radiation must not have been to more than 15% of marrow-producing locations.
11. Pregnant women are excluded from this study because the potential for teratogenic or abortifacient effects of AR-12 are not known. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with AR-12, breastfeeding should be discontinued if the mother is treated with AR-12.
12. Patients with known human immunodeficiency virus (HIV) are not eligible for this study.
13. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
14. Patients with QTc > 470 msec on Screening ECG or a clinically relevant ECG abnormality as determined by the investigator or his/her designee.
15. Patients with left bundle-branch block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study in adults with advanced or recurrent solid tumors or lymphoma is to evaluate the safety and tolerability of AR-12. | Every 2 Cycles (approximately 28 days per cycle)

SECONDARY OUTCOMES:
Evaluate PK samples during C1, identify and use biomarkers to characterize the PD effects in surrogate and tumor tissue, establish a biologically active dose range, assess preliminary anti-tumor activity in cancer patients. | C1 only in each dose cohort

CONTACTS AND LOCATIONS:
Overall Officials: James P Thomas, MD PhD, Principal Investigator — The Ohio State University Comprehensive Cancer Center; Raoul Tibes, MD PhD, Principal Investigator — TGen Clinical Research Services at Scottsdale Healthcare; Johann S de Bono, MD PhD, Principal Investigator — Royal Marsden Hospital - Drug Development Unit
Locations (3):
- United States (2):
  - TGen Clinical Research Services at Scottsdale Healthcare, Scottsdale, Arizona
  - The Ohio State University - Comprehensive Cancer Center, Columbus, Ohio
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom